CLINICAL TRIAL: NCT01680276
Title: Clinical and Cost Effectiveness of Staff Training in Positive Behaviour Support (PBS) for Treating Challenging Behaviour in People With Intellectual Disability: A Cluster Randomised Controlled Trial
Brief Title: Clinical and Cost Effectiveness of Positive Behaviour Support: a Trial
Acronym: PBS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/104/13
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2015-06

CONDITIONS: Challenging Behaviour
Keywords: intellectual disability; developmental disability; challenging behaviour; behavioural intervention; training
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PBS based staff training (Experimental): The training, which will be supported by a treatment manual will comprise the following sections:
  1. Functional Behavioural Assessment and formulation skills
     • Brief Behavioural Assessment Tool for brief functional analyses
  2. Primary Prevention
  3. Secondary Prevention and Reactive Strategies
  4. Periodic Service Review and Problem Solving
     * Developing individualised periodic service reviews
     * Trouble shooting
  Interventions: Behavioral: PBS based staff training; Other: Treatment as Usual
- Treatment as usual (Other): Most community intellectual disability services provide a range of health interventions that include but are not limited to psychiatric assessment and management, nursing support, psychology, speech and language therapy, occupational therapy and counselling. There may be some variation in resources but service users with challenging behaviour are likely to receive a range of broadly defined behavioural management and pharmacological interventions. Staff is routinely supervised by their clinical managers weekly.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: PBS based staff training — Please see published study protocol for more information:
  http://www.biomedcentral.com/1471-244X/14/219
  Arms: PBS based staff training
Other: Treatment as Usual — http://www.biomedcentral.com/1471-244X/14/219

SUMMARY:
Many people with intellectual disability have challenging behaviour which often has serious consequences such as the prescription of long term medication, in-patient admissions and disruption of normal daily activities. Community intellectual disability services may have difficulties in helping people with challenging behavior. Available research suggests that Positive Behavior Support (PBS), a training system that teaches staff how to manage these situations, can benefit service users who may show improvements in challenging behavior and quality of life. The investigators do not know of any study so far that has examined the clinical and cost effectiveness of PBS that is provided by staff in routine clinical practice in community intellectual disability services. If PBS proved to be better than treatment as usual, it would have important implications for the management of a very vulnerable group of service users. In this trial, health staff will receive accredited training in PBS available in a manual written by PBS experts. It will give details of how to understand challenging behavior and develop a management plan and how to implement it and monitor whether it has achieved its goals. Twenty community intellectual disability services and 260 service users with mild to severe intellectual disability and challenging behavior will be invited to take part in the study. The sample size calculations are based on our pilot study and allow for non participation of 10% and inflation due to the number of community intellectual disability teams and staff that will take part. The teams will be randomly allocated into one of two conditions. Half will be in the PBS arm (but will also have treatment as usual) and half will be in the treatment as usual only group. The investigators will carry out assessments of challenging behavior, use of services, quality of life, mental health, aggression and family and paid carer burden at six and 12 months. The investigators will monitor treatment fidelity and the investigators will talk to a sample of paid and family carers, service users, staff and managers about what they think of the treatment and how best the investigators can deliver it in routine care. The main outcome is reduction in challenging behavior at one year after the randomization. The investigators will also carry out a health economic evaluation to examine the costs and consequences of staff training in PBS.

DETAILED DESCRIPTION:
Please see published protocol at:

http://www.biomedcentral.com/1471-244X/14/219

ELIGIBILITY:
Inclusion Criteria:

* Service users: Eligible to receive care from intellectual disability services; mild to severe intellectual disability; aged 18 years and over; total ABC score of at least 15 (indicates a degree of challenging behaviour occurring at least weekly including verbal or physical aggression, hyperactivity, refusal to attend activities, non responsiveness that requires professional input).
* Service: Willing to participate; availability of at least two staff members willing to train; written agreement by the service manager to participate.

Exclusion Criteria:

* Service users: primary clinical diagnosis of personality disorder or substance misuse; relapse in pre-existing mental disorder; decision by clinical team that a referral to the study would be inappropriate, e.g. there is an open complaint investigation
* Service: there are no team members willing to train; the service has already received and implements accredited PBS for their service users.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Challenging Behaviour | 12 months
  Reduction in challenging behaviour as measured by the Aberrant Behaviour Checklist (ABC)and change from baseline and 6 months

SECONDARY OUTCOMES:
Quality of life | 12 months
  Improvement in Quality of Life measured by the Quality of Life Questionnaire
Mental health status | 12 months
  Improvement in mental health measured by the mini-PASADD.
Family carer burden | 12 months
  Reduction in family carer burden measured by the Uplift/Burden Scale
Paid carer burden | 12 months
  Reduction in burden measured by Caregiving Difficulty Scale-Intellectual Disability
Family Carer Psychiatric Morbidity | 12 months
  Reduction in Psychiatric morbidity measured by the General Health Questionnaire (12 item version)

OTHER OUTCOMES:
Cost effectiveness | 12 months
  Service use will be measured over the trial period at three month intervals using the Client Service Receipt Inventory adapted specifically for the study
Community participation | 6 months
  Improvement measured by change in Guernsey Community Participation and Leisure Activity Scale (GCPLAS)
Community participation | 12 months
  Positive change from 6 months as measured with the GCPLAS

CONTACTS AND LOCATIONS:
Overall Officials: Andre Strydom, MD PhD, Study Director — UCL; Ian Hall, MBBS MPhil, Study Director — East London Foundation Trust; Michael King, FRCGP PhD, Study Director — UCL; Rumana Omar, Study Director — UCL Statistics; Rachael Hunter, Study Director — Health Economist; Vivien Cooper, Study Director — Challenging Behaviour Foundation
Locations (3):
- United Kingdom (3):
  - Leicestershire Foundation Trust, Leicester
  - Camden & Islington Foundation Trust, London
  - South London and St George's Mental Health Trust, London

REFERENCES:
- [Background] Hassiotis A, Strydom A, Crawford M, Hall I, Omar R, Vickerstaff V, Hunter R, Crabtree J, Cooper V, Biswas A, Howie W, King M. Clinical and cost effectiveness of staff training in Positive Behaviour Support (PBS) for treating challenging behaviour in adults with intellectual disability: a cluster randomised controlled trial. BMC Psychiatry. 2014 Aug 3;14:219. doi: 10.1186/s12888-014-0219-6. PMID 25927187
- [Derived] Strydom A, Bosco A, Vickerstaff V, Hunter R; PBS study group; Hassiotis A. Clinical and cost effectiveness of staff training in the delivery of Positive Behaviour Support (PBS) for adults with intellectual disabilities, autism spectrum disorder and challenging behaviour - randomised trial. BMC Psychiatry. 2020 Apr 15;20(1):161. doi: 10.1186/s12888-020-02577-1. PMID 32293383
- [Derived] Hunter RM, Vickerstaff V, Poppe M, Strydom A, King M, Hall I, Crabtree J, Omar R, Cooper V, Biswas A, Hassiotis A. Staff training in positive behaviour support for behaviour that challenges in people with intellectual disability: cost-utility analysis of a cluster randomised controlled trial. BJPsych Open. 2020 Feb 5;6(2):e15. doi: 10.1192/bjo.2020.1. PMID 32019635
- [Derived] Hassiotis A, Poppe M, Strydom A, Vickerstaff V, Hall I, Crabtree J, Omar R, King M, Hunter R, Bosco A, Biswas A, Ratti V, Blickwedel J, Cooper V, Howie W, Crawford M. Positive behaviour support training for staff for treating challenging behaviour in people with intellectual disabilities: a cluster RCT. Health Technol Assess. 2018 Mar;22(15):1-110. doi: 10.3310/hta22150. PMID 29596045
- [Derived] Hassiotis A, Poppe M, Strydom A, Vickerstaff V, Hall IS, Crabtree J, Omar RZ, King M, Hunter R, Biswas A, Cooper V, Howie W, Crawford MJ. Clinical outcomes of staff training in positive behaviour support to reduce challenging behaviour in adults with intellectual disability: cluster randomised controlled trial. Br J Psychiatry. 2018 Mar;212(3):161-168. doi: 10.1192/bjp.2017.34. Epub 2018 Feb 12. PMID 29436314
- See also: Published protocol in open access journal — http://www.biomedcentral.com/1471-244X/14/219